CLINICAL TRIAL: NCT00497549
Title: Prospective Randomized Controlled Trial Comparing Side to Side Stapled and Hand Sewn Esophagogastric Anastomosis in the Neck
Brief Title: Trial Comparing Side-to-Side Stapled and Hand-sewn Esophagogastric Anastomosis in Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Sundeep Singh Saluja, Department of G I Surgery, AIIMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIS1/2004
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-04

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy; hand sewn anastomosis; side-to-side stapled
MeSH Terms: conditions — Esophageal Neoplasms | interventions — SAH-Bcl9

ARMS (2):
- 1 (Active Comparator): A proper site on the anterior wall of stomach away from the stapled line approximately 2 cm below the highest point of the gastric conduit will be anastamosed to esophagus Posterior interrupted seromuscular sutures will be taken with 3-0 silk. The stomach will then be opened transversely (2.5 to 3 cm long). Interrupted stitches with full thickness of the stomach and esophagus will be placed to achieve mucosa to mucosa approximation. A 16F nasogastric tube will then be placed across the anastomosis into the intrathoracic stomach. The anterior wall of the anastomosis will be completed in a manner similar to posterior wall.
  Interventions: Procedure: hand sewn
- 2 (Active Comparator): 5 cm of the mobilized stomach will be placed in the neck. Three interrupted sutures will be taken between the posterior wall of esophagus and anterior wall of stomach. A 1.5 cm gastrotomy will be made. Two stay sutures will then be taken, one at the anterior corner of esophagus and another between posterior corner of esophagus and the middle of the gastrotomy. The stapler device (Endopath, EZ45) will be introduced.The staple cartridge will then be rotated so that the posterior wall of the esophagus and the anterior wall of the stomach will align in a parallel manner and fire the stapler. A 16F nasogastric tube will be placed across the anastomosis and the anterior edges of the gastrotomy and open esophagus will be approximated with interrupted 3-0 silk.
  Interventions: Procedure: side-to-side stapled

INTERVENTIONS:
Procedure: side-to-side stapled — 5 cm of the mobilized stomach will be placed in the neck. Three interrupted sutures will be taken between the posterior wall of esophagus and anterior wall of stomach. A 1.5 cm gastrotomy will be made. Two stay sutures will then be taken, one at the anterior corner of esophagus and another between posterior corner of esophagus and the middle of the gastrotomy. The stapler device (Endopath, EZ45) will be introduced.The staple cartridge will then be rotated so that the posterior wall of the esophagus and the anterior wall of the stomach will align in a parallel manner and fire the stapler. A 16F nasogastric tube will be placed across the anastomosis and the anterior edges of the gastrotomy and open esophagus will be approximated with interrupted 3-0 silk.
  Other Names: stapled
  Arms: 2
Procedure: hand sewn — A proper site on the anterior wall of stomach away from the stapled line approximately 2 cm below the highest point of the gastric conduit will be anastamosed to esophagus Posterior interrupted seromuscular sutures will be taken with 3-0 silk. The stomach will then be opened transversely (2.5 to 3 cm long). Interrupted stitches with full thickness of the stomach and esophagus will be placed to achieve mucosa to mucosa approximation. A 16F nasogastric tube will then be placed across the anastomosis into the intrathoracic stomach. The anterior wall of the anastomosis will be completed in a manner similar to posterior wall.
  Arms: 1

SUMMARY:
Carcinoma esophagus is a common cause of dysphagia. Once dysphagia occurs, a majority of the tumours are advanced. Most of them would require some form of treatments for control of dysphagia and to improve the quality of life. Surgery is the only hope for cure. It requires complete removal of the esophagus. After removal of the esophagus, the stomach can be used as a substitute for the esophagus. Anastomosis can be done in the neck either by a hand-sewn or by a stapled anastomosis. The anastomotic leak rates reported in studies comparing hand-sewn with stapled anastomosis are variable. Many non-randomized studies have reported leak rate as low as 5% with stapled technique. However, the stricture rate is higher in the stapled group. There is no randomized study comparing hand-sewn anastomosis with side-to-side stapled anastomosis. Hence, the investigators planned a randomized trial comparing the anastomotic sequelae after hand-sewn anastomosis with stapled anastomosis in the neck.

DETAILED DESCRIPTION:
Hypothesis:

Side-to-side stapled anastomosis will decrease anastomotic leak rate by 15% compared to hand sewn technique in cervical esophagogastric anastomosis

Background:

Following esophagectomy or esophageal bypass, restoration of continuity by gastric interposition with cervical esophagogastric anastomosis (CEGA) can be done either by a hand-sewn or stapled anastomosis. Regardless of the surgical approach, decreasing anastomotic complications is essential for minimizing early morbidity and improving long-term functional results and quality of life. Cervical esophagogastric anastomosis almost eliminates the risk of postoperative mediastinitis associated with anastomotic leaks. Further, 98% of CEGA leaks can be managed successfully with local wound care (1), and less than 2% are associated with serious complications such as gastric tip necrosis, cervical vertebral osteomyelitis, epidural abscess and tracheogastroesophageal fistula, etc (2). Though early complications of CEGA are less, the long-term sequelae such as anastomotic stricture occur in nearly half the patients with an anastomotic leak. The need for life long esophageal dilatation negates the benefit of an operation intended to relieve dysphagia. The cause of anastomotic dehiscence in CEGA is possibly multifactorial (3,4) with both local tissue and systemic factors are being implicated. As the esophagus has no serosa, its longitudinal muscles hold sutures poorly and the awkward surgical exposure, possibly contribute to the higher anastomotic leak rates. Surgical technique is thus likely to play an important role. The incidence of CEGA leakage with hand sewn has been reported from 15% to 25% (5). While the stapled anastomosis is considered to be more expedient, less traumatic to tissues, with lower leak rates and associated with less mortality and morbidity, they are criticized for increased cost and high stricture rates. Most reports prior to 2000 showed identical leak rates in patients having a hand-sewn or stapled anastomosis with higher stricture rate in the stapled group (6-8). With recent technical refinements the CEGA has been performed in side-to-side manner using the Auto-Suture Endo-GIA 30-3.5 stapler. Following side to side anastomosis the leak rates have been reported to be less than 5%, with lower incidence of anastomotic stricture after leak and improved satisfaction in swallowing compared to hand sewn technique (9). These studies were retrospective and demanded a randomized trial to confirm the results. We therefore planned a randomized trial comparing the anastomotic sequelae after hand-sewn anastomosis with mechanical stapled side-to-side anastomosis

Objective:

To compare the rates of anastomotic leaks and postoperative benign stricture after CEGA done by hand-sewn (end-to-side) technique or by linear stapled anastomosis (side-to-side) technique.

PATIENTS AND METHODS:

All the patients who attended outpatient department of GI Surgery with complaints of dysphagia will be evaluated for esophageal disorder. After confirming the diagnosis of esophageal cancer and decision of esophagectomy, patients will be included in our study.

Inclusion criteria i Any patient with resectable carcinoma of the mid or lower thoracic esophagus and gastro-esophageal junction. ii Benign esophageal lesion where esophageal resection was beneficial and feasible.

Exclusion criteria i Patients who had upper thoracic or cervical esophageal carcinoma ii Unresectable lesions (T4/M1) iii Prior gastric surgery iv Poor performance status (ECOG 3,4) Sample size calculation The number of patients to be included was calculated to be 87 patients in each group based on the assumption that anastomotic leak rate will be reduced to 5% using side-to-side stapled anastomosis. The sample size was calculated by the formula for a power of 80% and alpha error of 0.05.

They will be randomly divided into two groups using computer generated random numbers.

Group A Hand sewn anastomosis; Group B Stapled anastomosis Written informed consent will be obtained from each patient before entry into the study.

Diagnostic work up and preoperative preparation The diagnostic work-up will include barium swallow, upper gastrointestinal (UGI) endoscopy and biopsy (where malignancy was suspected), hypopharyngoscopy (for corrosive stricture of esophagus), as well as haemogram, serum chemistry, liver function tests, ECG, chest x-ray and pulmonary function tests. In the malignant group, preoperative imaging will also include computed tomography (CT) scan from the neck to the upper abdomen including the liver and celiac axis. Preoperative nutrition will be maintained and if required a ryle tube or feeding jejunostomy will be done. Incentive spirometry, steam inhalation, bronchodilators and antibiotics will be used to improve the pulmonary status as required.

At surgery, the operative procedures, time taken for anastomosis and total operating time will be recorded. After surgery, patients will be assessed for anastomotic leakage by a radiographic contrast (gastrografin) study to be performed on seventh postoperative day. Anastomotic leakage will be defined as a radiological defect at the anastomotic site or leakage of swallowed fluid out of the drain site or cervical wound. Other complications, including cardiopulmonary morbidity, septic complications, duration of hospital stay after surgery and operative mortality will also be studied. Operative mortality included all patients who will die within 30 days of the procedure or during the same hospital admission. Anastomotic stricture will be defined as failure to pass the esophagoscope through the anastomosis or anastomotic narrowing requiring dilatation to relieve dysphagia.

Surgical technique:

The surgical approach will be either transhiatal or transthoracic esophagectomy. The gastric conduit will be prepared based on the right gastric and right gastroepiploic vessels and pyloromyotomy and pyloroplasty will not performed except in patients with corrosive strictures. Finger dilatation of pylorus will be done when required. The conduit will be prepared using 75-mm linear cutter. The stomach will be brought up into the neck through either the retrosternal or posterior mediastinal route. The CEGA will be done by a side-to-side stapled or end-to-side hand-sewn method. Chest tubes (32F) will be inserted bilaterally to take care of any breach in the pleura. Feeding jejunostomy (Witzel's type) with 12F Malecot's catheter will be done in all patients. The neck wound will be closed loosely with interrupted 3-0 vicryl sutures over a 14F suction drain and the skin will be approximated with skin staplers.

Hand-sewn anastomosis: A proper site on the anterior wall of stomach away from the stapled line approximately 2 cm below the highest point of the gastric conduit will be anastamosed to esophagus Posterior interrupted seromuscular sutures will be taken with 3-0 silk. The stomach will then be opened transversely (2.5 to 3 cm long). Interrupted stitches with full thickness of the stomach and esophagus will be placed to achieve mucosa to mucosa approximation. A 16F nasogastric tube will then be placed across the anastomosis into the intrathoracic stomach. The anterior wall of the anastomosis will be completed in a manner similar to posterior wall.

Stapled anastomosis: At least 5 cm of the mobilized stomach will be placed in the neck. Three interrupted seromuscular sutures will be taken between the posterior wall of the esophagus and anterior wall of stomach well away from the gastric staple line. A 1.5 cm gastrotomy will be made. Two stay sutures will then be taken, one at the anterior corner of the esophagus and another between the posterior corner of esophagus and the middle of the gastrotomy. These stay sutures will be retracted downwards as the stapler device (using Endopath, EZ45 Endoscopic Linear Cutter) will be introduced, the thinner portion into the stomach and the thicker staple-bearing portion into the esophagus. The staple cartridge will then be rotated so that the posterior wall of the esophagus and the anterior wall of the stomach will align in a parallel manner, keeping the site of the anastomosis well away from the gastric staple suture line and fire the stapler. A 16F nasogastric tube will be placed across the anastomosis into the intrathoracic stomach, and the anterior edges of the gastrotomy and open esophagus will be approximated in two layers with interrupted 3-0 silk.

Postoperative management: The nasogastric tube will be removed on the 3rd postoperative day. Jejunostomy trial feed will be started intestinal activity will appear. If there is no obvious leak, bedside test feeding with water will be done on the 5th postoperative day. If bedside test feeding shows no leak, oral feeding will be started gradually with water, banana, curds and soft diet. A contrast study will be done on the 7th postoperative day unless there is an obvious anastomotic leak. The neck drain will be removed after the contrast study. If a leak is identified, the cervical wound will be opened to establish external drainage of any cervical abscess and anastomotic fistulae. Regular dressing with normal saline soaked gauze will be done. If there is no clinical leak but the contrast study shows a contained leak (type 1 leak), patients will be managed conservatively without opening the cervical wound.

Follow up:

All patients will be followed one week after discharge and at 3-month intervals for the first two years. Routine clinical examination, hemogram and liver function tests will be done in all patients. Dysphagia will be assessed with barium swallow and esophagoscopy. Anastomotic strictures will be dilated with endoscopic or by a Foley catheter balloon (This technique has been adapted for home based self dilatation) (10).

Statistical analysis:

Continuous variables will be reported as Mean with Standard Error of Mean (SEM). Categorical variables will be reported as proportions. Student's t test, Chi-square tests and Fisher's exact test where appropriate will be used for comparison between groups. A p value of 0.05 or less will be regarded as significant.

REFERENCES

1. Orringer MB, Lemmer JH. Early dilation in the treatment of esophageal disruption. Ann Thorac Surg 1986;42:536-9
2. Iannettoni MD, Whyte RI, Orringer MB. Catastrophic complications of the cervical esophagogastric anastomosis. J Thorac Cardiovasc Surg 1995;110:1493-1501
3. Dewar L, Gelfand G, Finley RJ, Evans K, Inculet R, Nelems B. Factors affecting cervical anastomotic leak and stricture formation following esophagogastrectomy and gastric tube interposition. Am J Surg 1992;163:484-9
4. Gupta NM, Gupta R, Rao MS, Gupta V. Minimizing cervical esophageal anastomotic complications by a modified technique. Am J Surg 2001;181:534-9
5. Orringer MB, Marshall B, Iannettoni MD. Transhiatal esophagectomy: clinical experience and refinements. Ann Surg 1999;230:392-403
6. Fok M, Ah-Chong AK, Cheng SW, Wong J. Comparison of a single layer continuous hand-sewn method and circular stapling in 580 oesophageal anastomosis. Br J Surg 1991;78:342-5
7. Law S, Fok M, Chu KM, Wong J. Comparison of hand-sewn and stapled esophagogastric anastomosis after esophageal resection for cancer: a prospective randomized controlled trial. Ann Surg 1997;226:169-73
8. Beitler AL, Urschel JD. Comparison of stapled and hand-sewn esophagogastric anastomoses. Am J Surg 1998;175:337-40
9. Orringer MB, Marshall B, Iannettoni MD. Eliminating the cervical esophagogastric anastomotic leak with a side-to-side stapled anastomosis. J Thorac Cardiovasc Surg 2000;119:277-88
10. Shad SK, Gupta S, Chattopadhyay T Self-dilatation of cervical oesophagogastric anastomotic stricture: a simple and effective technique. Br J Surg 1991;78:1254-5

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with resectable carcinoma of the mid or lower thoracic esophagus and gastroesophageal junction
2. Benign esophageal lesion where esophageal resection was beneficial and feasible

Exclusion Criteria:

1. Patients who had upper thoracic or cervical esophageal carcinoma
2. Irresectable lesions (T4/M1)
3. Prior gastric surgery
4. Poor performance status

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-07; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage defined as a radiological defect at the anastomotic site or leakage of swallowed fluid out of the drain site or cervical wound. | within 7 days
  It was defined as a radiological defect at the anastomotic site or leakage of swallowed fluid out of the drain site or cervical wound

CONTACTS AND LOCATIONS:
Overall Officials: Tushar K Chattopadhyay, MS, Study Director — Deptt. GI Surgery, All India Institute of Medical sciences, New Delhi, India; Sundeep S Saluja, MS, MCh, Principal Investigator — Deptt. GI Surgery, All India Institute of Medical sciences, New Delhi, India
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Law S, Fok M, Chu KM, Wong J. Comparison of hand-sewn and stapled esophagogastric anastomosis after esophageal resection for cancer: a prospective randomized controlled trial. Ann Surg. 1997 Aug;226(2):169-73. doi: 10.1097/00000658-199708000-00008. PMID 9296510
- [Background] Orringer MB, Marshall B, Iannettoni MD. Eliminating the cervical esophagogastric anastomotic leak with a side-to-side stapled anastomosis. J Thorac Cardiovasc Surg. 2000 Feb;119(2):277-88. doi: 10.1016/S0022-5223(00)70183-8. PMID 10649203
- [Derived] Saluja SS, Ray S, Pal S, Sanyal S, Agrawal N, Dash NR, Sahni P, Chattopadhyay TK. Randomized trial comparing side-to-side stapled and hand-sewn esophagogastric anastomosis in neck. J Gastrointest Surg. 2012 Jul;16(7):1287-95. doi: 10.1007/s11605-012-1885-7. Epub 2012 Apr 24. PMID 22528571